CLINICAL TRIAL: NCT04458779
Title: Cardiovascular Effects of Continuous Positive Airway Pressure in Patients With Acute Stroke and Obstructive Sleep Apnea
Brief Title: Continuous Positive Airway Pressure on Acute Stroke and Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chou-Han Lin, Principical investigator, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109018-E
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Stroke, Acute; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; stroke; continuous positive airway pressure
MeSH Terms: conditions — Stroke; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP group (Experimental): Subjects will receive CPAP treatment in addition to optimal standard therapy for acute stroke.
  Interventions: Device: CPAP
- Usual-care group (No Intervention): Subjects will receive optimal standard therapy for acute stroke.

INTERVENTIONS:
Device: CPAP — CPAP will be given after obstructive sleep apnea being diagnosed in the acute stage of stroke.
  Arms: CPAP group

SUMMARY:
Stroke affects 16.9 million individuals each year and is the second leading cause of death worldwide. Despite advances in pharmacologic therapy, morbidity , mortality and rates of hospitalization for stroke remain high. These data emphasize the importance of identifying all treatable conditions that could aggravate stroke. One such condition is obstructive sleep apnea (OSA).

Sleep-related breathing disorders, including obstructive and central sleep apnea, often coexist with stroke. Compared to the general population, in whom OSA is the most common form of this breathing disorder with recent prevalence estimates of 22% of male and 17% of female , in the stroke population, the prevalence of OSA is much greater at 70% . Several randomized controlledtrials on OSA patients with stroke in acute or sub-acute stage showed that treating OSA with continuous positive airway pressure (CPAP) improved motor and functional outcomes, accelerated neurological recovery.Apart from the benefits in better neurological outcomes, secondary analyses of SAVE study suggested that CPAP treatment potentially help to reduce recurrence of stroke. Nevertheless, we don't have evidence yet from randomized control studies to prove CPAP treatment would reduce the recurrence of cardiovascular or cerebrovascular events.

Traditionally, recurrence of cardiovascular or cerebrovascular events uses documented mortality, morbidity or hospitalization for heart failure, acute coronary syndrome or stroke as clinical endpoints. Recently, several studies showed that enlarged left atrium (LA) can serve as a predictor for recurrent stroke or cardiovascular events. On the other hand, a growing body of studies demonstrated that CPAP treatment reduce size of LA in those with OSA. Notably, all of these studies above are observational or retrospective in nature. To date, there are no prospective longitudinal randomized controlled trials reporting the effect of CPAP treatment of OSA on the change of size of LA. We therefore will undertake a randomized , controlled trial involving patients with stroke to test the primary hypothesis that treatment of OSA with CPAP would reduce the size of LA.

ELIGIBILITY:
Inclusion Criteria:

1. Time from onset of stroke symptoms to hospital arrival <2 weeks .
2. Stroke is documented with brain magnetic imaging or computed tomography
3. Competency to provide informed consent.
4. Moderate to severe obstructive sleep apnea being established with the use of a home sleep-study screening device (ApneaLink).
5. Epworth sleepiness scale≦10.

Exclusion Criteria:

1. Having received CPAP for obstructive sleep apnea prior to admission.
2. History of pneumothorax or brain surgery.
3. Coexisting heart failure or renal failure or persistent atrial fibrillation.
4. Unable to wear a nasal or nasal-oral mask.
5. Concomitant uncontrolled infection.
6. Swallowing difficulty or episodes of choking due to stroke
7. Coexisting central nervous diseases such as dementia

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in left atrium volume index (LAVI) | 12 months
  Change of LAVI will be assessed by transthoracic echocardiography at baseline and at 3, 6 and 12 months post randomization.
Serial change of NT-proBNP | 12 months
  Change of NT-proBNP will be assessed at baseline and at 3, 6 and 12 months post randomization.

SECONDARY OUTCOMES:
Neurological and functional assessments-1 | 12 months
  Change in National Institutes of Health (NIH) stoke scale will be assessed at baseline ,3, 6 and 12 months post randomization.
Neurological and functional assessments-2 | 12 months
  Change in modified Rankin scale will be assessed at baseline, 3, 6 and 12 months post randomization.
Neurological and functional assessments-3 | 12 months
  Chang in Barthel-ADL index will be assessed at baseline, 3, 6 and 12 months post randomization.
Change in Quality of life assessments | 12 months
  Change in Epworth sleepiness scale and Medical Outcomes Study 36-Item Short-Form Health Survey at baseline, 3, 6 and 12 months post randomization.

OTHER OUTCOMES:
Numbers of cardiovascular or cerebrovascular events | 12 months
  Numbers of cardiovascular or cerebrovascular events post randomization
Time to cardiovascular or cerebrovascular events | 12 months
  Time to cardiovascular or cerebrovascular events post randomization
Numbers of all-cause hospitalizations | 12 months
  Numbers of hospitalizations for any reason post randomization
Number of deaths | 12 months
  Numbers of deaths from all causes post randomization
Time to deaths | 12 months
  Time to deaths from all causes post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Chou-Han Lin, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan